CLINICAL TRIAL: NCT00637884
Title: A Single-Center, Randomized, Double-Blind, Placebo-Controlled, Two-Way Crossover Study Designed to Evaluate the Efficacy of Fexofenadine HCl 180 mg for Preventing and Controlling Cat Allergy Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M016455A_4148
Record Dates: First submitted 2008-03-10; First posted 2008-03-18 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Cat Induced Allergic Rhinitis
MeSH Terms: interventions — fexofenadine

INTERVENTIONS:
Drug: Fexofenadine HCl

SUMMARY:
This is a single-center, prospective, randomized, double-blind, placebo-controlled, two-way crossover study. A live cat challenge model will be used for exposing subjects to Fel d1. Subjects who test positive for cat allergy symptoms during a priming cat exposure challenge will be eligible to enter the treatment phase of the study. Baseline efficacy measures will be obtained prior to the dispensing of study medication during both treatment periods. Cat challenges will be initiated 1.5 hours following treatment with study medication.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, aged 12 years and older, inclusive
* History of cat-induced allergic rhinitis for at least 2 years, requiring the use of allergy medication or resulting in avoidance of cats
* Skin test positive to cat allergen at screening, defined as a wheal greater than one-half the diameter of the histamine control and at least 3 mm larger than the diameter of the glycerin-saline solution control. A skin test performed in the previous 15 months may be used to qualify the subject if it was performed at the investigator's site and recorded in the subject's medical record
* FEV1 greater than or equal to 80% of the predicted value on the screening assessment, and at the baseline assessment prior to the priming cat challenge(s). After the priming cat challenge, FEV1 must not have decreased >12% from the pre-challenge testing % predicted value
* Reversibility of <12% in absolute FEV1 following 2 puffs of albuterol at screening
* Minimal baseline allergic symptoms, defined as TSS less than or equal to 4 at the baseline assessments prior to the priming cat challenges
* All females must have a negative urine pregnancy test
* Willing and able to adhere to visit schedules and all study requirements
* Mild to moderate allergic symptoms defined as TSS less than or equal to 8 at screening

Exclusion Criteria:

* Asthma that requires treatment with medication other than inhaled, short-acting beta-agonists (not to be taken within 6 hours prior to the priming visit(s) or Visits 3 or 4) or asthma known to be exacerbated by exposure to Fel d1. (Subjects with exercise-induced asthma will be allowed.)
* Requires medication for rhinitis that cannot be withheld
* Has a cat in the home (Subjects who have cats who are exclusively outdoors will be allowed.)
* Upper respiratory infection within 4 weeks of study entry
* History of severe reactions to cat exposure by self-report (severe is defined as being unable to tolerate cat exposure for at least 30 minutes)
* Acute or chronic sinusitis or other nasal diseases that resulted in nasal obstruction (e.g., nasal septum deviation, nasal polyps) within 4 weeks of study entry
* Known hypersensitivity to fexofenadine HCl or to drugs with similar chemical structures
* Clinically significant ECG values that, in the judgment of the investigator, would have clinical implications for the subject's participation in the study
* Clinically significant medical condition (such as cardiovascular, hepatic, neurologic, hematological, renal, gastrointestinal, endocrine, or other major systemic disease), that, in the judgment of the investigator, might interfere with the study, require treatment or make implementation of the protocol or interpretation of the study results difficult
* Pregnant or breast-feeding
* Likely to require treatment during the study period with drugs not permitted by the study protocol
* Immunotherapy, except those on a constant dose of immunotherapy that will be maintained throughout the study
* Treatment with an investigational agent or device within 30 days prior to study entry
* Recent history of alcohol or other drug abuse
* Mental condition that renders the subject unable to understand the nature, scope, and possible consequences of the study
* Unlikely to comply with the protocol (e.g., has an uncooperative attitude, is unlikely to complete the study)
* Subjects who are research employees or relatives of study site staff involved in this study or those who have or will read the protocol

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2003-11; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Determine efficacy of fexofenadine HCl 180 mg versus placebo in preventing and controlling self-reported cat allergy symptoms in subjects who have a known allergy to cats and who are exposed to feline domesticus allergen 1

SECONDARY OUTCOMES:
Determine efficacy of fexofenadine HCl 180 mg compared to placebo in subjects with a known allergy to cats

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, Study Director — Sanofi